CLINICAL TRIAL: NCT03711877
Title: Comparative Study of Scalp Cooling System and Chemical Cold Cap on Prevention of Chemotherapy-induced Alopecia in Women With Breast Cancer
Brief Title: Comparative Study of Scalp Cooling System and Chemical Cold Cap (COHAIR Study)
Acronym: COHAIR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tao OUYANG (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Director of Breast Center of Peking University Cancer Hospital, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BCP-25
Record Dates: First submitted 2018-10-11; First posted 2018-10-19 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Primary Breast Cancer
Keywords: alopecia; scalp cooling system; cold cap
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scalp cooling system (Experimental): 'Scalp cooling device' will be used to prevent alopecia during chemotherapy regimen infusion.
  Interventions: Device: Scalp cooling system
- cold cap (Active Comparator): 'Cold cap' will be used to prevent alopecia during chemotherapy regimen infusion.
  Interventions: Device: Cold cap

INTERVENTIONS:
Device: Scalp cooling system — Scalp cooling was initiated 30 minutes prior to each chemotherapy cycle, with scalp temperature maintained at 3°C (37°F) throughout chemotherapy and for 90 minutes to 120 minutes afterward. Temperature of scalp cooling system can be controlled constantly, the effect of reducing scalp temperature maybe better and patient tolerance maybe better. Meanwhile, there is a higher likelihood of hair retention due to a tight fit in scalp cooling system.
  Other Names: DigniCap
  Arms: scalp cooling system
Device: Cold cap — The operation of chemical cold cap is convenient and the price was low, and the economic burden of patients was not increased. But it is necessary to replace the cold cap periodically during chemotherapy, and the temperature during chemotherapy is difficult to keep constant.
  Arms: cold cap

SUMMARY:
This is a phase III, single-center, prospective, open-label, randomized,controlled study

DETAILED DESCRIPTION:
To conduct a prospective randomized controlled study comparing the effect of scalp cooling system (DigniCap) and chemical cold cap on preventing chemotherapy-induced alopecia in a group of breast cancer patients receiving standard anthracycline followed paclitaxel regimens. To obtain the exact data on the role of different methods of preventing alopecia in Chinese women with breast cancer.

PASS 11 software was used to calculate the sample size. According to the results of previous studies, the hair retention rate of the cold cap group was 67.7%, the hair retention rate of the scalp cooling system group was 50.5%, α=0.05，Power=0.8. The sample size was calculated to be at least 128 cases in each group, 256 cases in total.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 18≦age ≦66 years
* Invasive breast cancer diagnosed with core needle needle biopsy
* Staging I-II
* Without chemotherapy contraindications, and planned to receive neoadjuvant chemotherapy with a standard regimen (containing 4-cycle dose-dense anthracycline followed 4-cycle paclitaxel)
* Attend the study voluntarily, sign the informed consent

Exclusion Criteria:

* History of malignant tumors
* With chemotherapy contraindications
* With severe dermatosis and severe sparsity
* History of chronic diseases such as cerebrovascular disease, migraine and hyperthyroidism
* Uncontrolled diseases(e.g., heart failure, myocardial infarction within 6 months, arrhythmia, unstable diabetes, hypercalcemia) or active infection
* Refuse to join the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The effects on the prevention of alopecia of two methods | One year after neoadjuvant chemotherapy
  To compare the effects of scalp cooling system and chemical cold cap on the prevention of chemotherapy-induced alopecia in breast cancer patients undergoing neoadjuvant chemotherapy containing anthracycline followed paclitaxel. To assess hair status, a total of three photographs of patients'hair in the both groups were taken by study personnel before the start of first chemotherapy cycle, within 2 days before the start of paclitaxel chemotherapy and within 1 week after the last chemotherapy cycle. Photographs captured hair from the top of head. Patients assessed and estimated the percentage of hair loss using WHO classification of acute and subacute toxicity of anticancer drugs. Success was defined as WHO criteria alopecia grade I (<25% hair loss) or grade II (25%-50% hair loss). Failure was defined as WHO criteria alopecia grade III (>50% hair loss) or grade IV. The primary efficacy end point was assessed by clinicians who were independent.

SECONDARY OUTCOMES:
Qualify of life | One year after neoadjuvant chemotherapy
  To compare the effects of scalp cooling system and chemical cold cap on the quality of life. Quality of life was measured using the European Organization for Research and Treatment of Cancer Breast CancerSpecific Quality of Life Questionnaire-Core 30（EORTC QLQ-C30） administered at baseline and at the time of the last chemotherapy cycle.
Psychological stress | One year after neoadjuvant chemotherapy
  The Hospital Anxiety and Depression Scale (HADS) administered at baseline and at the time of the last chemotherapy cycle was used to assess anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Yu, Master, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China